CLINICAL TRIAL: NCT01570283
Title: ARMS - Administration Of Rapidly Generated Multivirus-Specific Cytotoxic T-Lymphocytes For The Prophylaxis And Treatment Of EBV, CMV, Adenovirus, HHV6, And BK Virus Infections Post Allogeneic Stem Cell Transplant
Brief Title: ARMS - Rapidly Generated Multivirus-Specific CTLs for Prophylaxis & Treatment of EBV, CMV, Adenovirus, HHV6 & BK Virus
Acronym: ARMS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AlloVir (Industry)
Collaborators: Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-29966 ARMS
Record Dates: First submitted 2012-03-27; First posted 2012-04-04 (Estimated); Results first posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-04

CONDITIONS: Viral Infection
Keywords: post allogeneic hematopoietic stem cell transplant; cytotoxic T lymphocytes; Cytomegalovirus; CMV; adenovirus; Epstein-Barr virus; EBV; Human polyomavirus type I; BK virus; Human herpesvirus 6; HHV6
MeSH Terms: conditions — Virus Diseases; Adenoviridae Infections; Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Multivirus-specific T cells 5*10^6 mCTLs/m2 for Prophylaxis (Experimental): Cohort 1 prophylaxis: Participants were administrated 5*10^6 mCTLs/m multivirusspecific T cells intravenously for prophylaxis of EBV, CMV, Adenovirus, HHV6 and BK virus infections post allogeneic stem cell transplant.
  Interventions: Biological: Multivirus-specific T cells Dose Level 1
- Multivirus-specific T cells 5*10^6 mCTLs/m2 for Treatment (Experimental): Cohort 1 treatment: Participants were administrated 5*10^6 mCTLs/m multivirusspecific T cells intravenously for treatment of EBV, CMV, Adenovirus, HHV6 and BK virus infections post allogeneic stem cell transplant.
  Interventions: Biological: Multivirus-specific T cells Dose Level 1
- Multivirus-specific T cells 1*10^7 mCTLs/m2 for Prophylaxis (Experimental): Cohort 2 prophylaxis: Participants were administrated 1*10^7 mCTLs/m multivirusspecific T cells intravenously for prophylaxis of EBV, CMV, Adenovirus, HHV6 and BK virus infections post allogeneic stem cell transplant.
  Interventions: Biological: Multivirus-specific T cells Dose Level 2
- Multivirus-specific T cells 1*10^7 mCTLs/m2 for Treatment (Experimental): Cohort 2 treatment: Participants were administrated 1*10^7 mCTLs/m multivirusspecific T cells intravenously for treatment of EBV, CMV, Adenovirus, HHV6 and BK virus infections post allogeneic stem cell transplant.
  Interventions: Biological: Multivirus-specific T cells Dose Level 2
- Multivirus-specific T Cells 2*10^7 mCTLs/m2 for Prophylaxis (Experimental): Cohort 3 prophylaxis: Participants were administrated 2*10^7 mCTLs/m multivirusspecific T cells intravenously for prophylaxis of EBV, CMV, Adenovirus, HHV6 and BK virus infections post allogeneic stem cell transplant.
  Interventions: Biological: Multivirus-specific T cells Dose Level 3
- Multivirus-specific T Cells 2*10^7 mCTLs/m2 for Treatment (Experimental): Cohort 3 treatment: Participants were administrated 2*10^7 mCTLs/m multivirusspecific T cells intravenously for treatment of EBV, CMV, Adenovirus, HHV6 and BK virus infections post allogeneic stem cell transplant.
  Interventions: Biological: Multivirus-specific T cells Dose Level 3

INTERVENTIONS:
Biological: Multivirus-specific T cells Dose Level 1 — The feasibility and safety of 3 different dose levels will be evaluated and will determine the maximum tolerated dose (MTD) level.
  Dose Level One: 5x10^6 mCTLs/m2
  There may be an option of administering 2 additional doses (at the same level the patient was receiving), 28 days after the first dose, in subjects that have a partial response after one dose or who receive other therapy that may affect the persistence or function of the infused CTL.
  Arms: Multivirus-specific T cells 5*10^6 mCTLs/m2 for Prophylaxis; Multivirus-specific T cells 5*10^6 mCTLs/m2 for Treatment
Biological: Multivirus-specific T cells Dose Level 2 — The feasibility and safety of 3 different dose levels will be evaluated and will determine the maximum tolerated dose (MTD) level.
  Dose Level Two: 1x10^7 mCTLs/m2
  There may be an option of administering 2 additional doses (at the same level the patient was receiving), 28 days after the first dose, in subjects that have a partial response after one dose or who receive other therapy that may affect the persistence or function of the infused CTL
  Arms: Multivirus-specific T cells 1*10^7 mCTLs/m2 for Prophylaxis; Multivirus-specific T cells 1*10^7 mCTLs/m2 for Treatment
Biological: Multivirus-specific T cells Dose Level 3 — The feasibility and safety of 3 different dose levels will be evaluated and will determine the maximum tolerated dose (MTD) level.
  Dose Level Three: 2x10^7 mCTLs/m2
  There may be an option of administering 2 additional doses (at the same level the patient was receiving), 28 days after the first dose, in subjects that have a partial response after one dose or who receive other therapy that may affect the persistence or function of the infused CTL
  Arms: Multivirus-specific T Cells 2*10^7 mCTLs/m2 for Prophylaxis; Multivirus-specific T Cells 2*10^7 mCTLs/m2 for Treatment

SUMMARY:
The subjects eligible for this trial have a type of blood cell cancer, other blood disease or a genetic disease for which they will receive a stem cell transplant. The donor of the stem cells will be either the subject's brother or sister, or another relative, or a closely matched unrelated donor. The Investigators are asking subjects to participate in this study which tests if blood cells from the subject's donor that have been grown in a special way, can prevent or be a effective treatment for early infection by five viruses - Epstein Barr virus (EBV), cytomegalovirus (CMV), adenovirus, BK virus (BKV) and human herpes virus 6 (HHV6).

The Investigators have grown T cells from the subject's stem cell donor in the laboratory in a way that will train them to recognize the viruses and control them when the T cells are given after a transplant. This treatment with specially trained T cells (also called cytotoxic T cells or "CTLs") has had activity against three of these viruses (CMV, EBV and Adenovirus) in previous studies. In this study the Investigators want to see if they increase the number of viruses that can be targeted to include BKV and HHV6 using a simple and fast approach to make the cells.

The Investigators want to see if they can use a kind of white blood cell called T lymphocytes (or T cells) to prevent and treat adenovirus, CMV, EBV, BKV and HHV6 in the early stages of reactivation or infection.

DETAILED DESCRIPTION:
To make the CTLs, subject's donors' cells were mixed with small pieces of proteins, called peptides that come from adenovirus, CMV, EBV, BKV and HHV6. These peptides stimulate donor T cells that react against the viruses to grow and train the donor T cells to kill cells that are infected with CMV, EBV, adenovirus, BKV and HHV6. Once sufficient numbers of T cells were made, they were tested to make sure they would target the cells infected with these viruses but not the normal cells. Then the cells were frozen.

When the Investigators think the subject needs them, the subject's donor's CTL cells will be thawed and injected into the intravenous line. To prevent an allergic reaction, prior to receiving the CTLs the subject may be given diphenhydramine (Benadryl) and acetaminophen (Tylenol). After the subject receives the cells, Investigators will monitor the levels of these five viruses in the blood. They will also take blood to see how long the T cells they gave the subject are lasting in the body.

If the CTL infusion has helped the subjects infection or if they have had a treatment, for example with steroid drugs that might have destroyed the T cells the subject was given, then they are allowed to receive up to 2 more doses of the cells.

The first part of this study was a dose escalation study. That means that at the beginning, patients were started on the lowest dose (1 of 3 different levels) of T cells. The next group of patients were started at a higher dose. This process continued until all 3 dose levels were studied. They would now like to enroll more patients at the highest dose level to get more information about how the T cells work.

Subjects will continue to be followed by their transplant doctors after the injection. The subject will either be seen in the clinic or they will be contacted by a research nurse to follow up for this study every week for 6 weeks then at 8 week and 3, 6 and 12 months. The subject may have other visits for their standard care. Subjects will also have regular blood tests done to follow their counts and the viral infection. To learn more about the way the T cells are working in the body, up to an extra 30-40 ml (6-8 teaspoons) of blood will be taken before the infusion and then at 1, 2, 4, 5, 6 and 8 weeks and 3 months. Blood should come from the central intravenous line, and should not require extra needle sticks.

If subjects experience a positive response or are taking medicines (such as steroids) that may affect how long T cells stay in the body, they may be able to receive up to two additional doses of the T cells at the same initial dose level from 28 days after their initial dose. After each T-cell infusion, they will be monitored as described above.

Study Duration: Subjects will be on study for approximately one year. If they receive additional doses of the T cells as described above, they will be followed until 1 year after their last dose of T-cells.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible following any type of allogeneic transplant to receive CTLs as prevention or for early reactivations as defined below.

1. Prior myeloablative or non-myeloablative allogeneic hematopoietic stem cell transplant using either bone marrow or peripheral blood stem cells within 12 months.
2. Prevention for patients at risk of CMV, adenovirus, EBV, BK virus, or HHV6 infection
3. Treatment of reactivation or infection which is defined for each virus as below

   * CMV- CMV antigenemia is monitored at least weekly post transplant. Reactivation is defined at CMV antigenemia with <10 leukocytes positive or elevated PCR. If any patient develops CMV antigenemia with >10 leukocytes positive or clinical evidence of CMV infection (defined as the demonstration of CMV by biopsy specimen from visceral sites (by culture or histology) either pre or after CTL infusions, standard treatment with Ganciclovir, and/or Foscarnet and Immunoglobulins will be initiated. Patients may receive CTLs for antigenemia or elevated PCR without visceral infection.
   * Adenovirus- Adenovirus infection will be defined as the presence of adenoviral positivity as detected by PCR or culture from ONE site such as stool or blood or urine or nasopharynx.

   Adenovirus disease will be defined as the presence of adenoviral positivity as detected by culture from more than two sites such as stool or blood or urine or nasopharynx.

   In patients who meet the criteria for disease Cidofovir may be added unless the subject could not tolerate this agent due to nephrotoxicity. Patients may receive CTLs for elevated PCR in blood or stool.
   * EBV- EBV-LPD is defined according to recent guidelines as proven EBV-LPD defined by biopsy or probable EBV-LPD defined as an elevated EBV DNA level associated with clinical symptoms (adenopathy or fever or masses on imaging) but without biopsy confirmation. Patients with EBV DNA reactivation only may receive CTLs on study. Patients with proven or probable EBV-LPD should also receive Rituxan
   * BK virus- Patients post transplant may develop asymptomatic BKV viruria or viremia. BK reactivation will be defined as detection of elevated BK levels by PCR in blood or urine while disease will be defined as detection in multiple sites or in one site with symptoms. Cidofovir has been administered intravenously in a low dose (i.e. up to 1 mg/kg 3 times weekly, without probenecid) or a high dose (ie, 5 mg/kg per week with probenecid) to HSCT patients with BK infections but no randomized trials are available proving its clinical efficacy. In patients who meet the criteria for disease Cidofovir may be added unless the subject could not tolerate this agent due to nephrotoxicity.
   * HHV6- HHV6 reactivation will be defined as detection of elevated HHV6 levels by PCR in blood while disease will be defined as detection in multiple sites or in one site with symptoms. Ganciclovir, Cidofovir, and foscarnet have variable in vitro activity against HHV-6, and may have a role in treating HHV-6-associated disease - hence one or more of these agents will be added in patients with disease.
4. Treatment may be given to eligible patients with a single or multiple infections. Patients with multiple infections with one or more reactivation and one or more controlled infection are eligible to enroll.
5. Clinical status at enrollment to allow tapering of steroids to less than 0.5 mg/kg/day prednisone.
6. Karnofsky/Lansky score of ≥ 50
7. ANC greater than 500/µL.
8. Bilirubin </= 2x upper limit normal
9. AST </= 3 x upper limit normal
10. Serum creatinine </= 2 x upper limit normal
11. HgB > 8.0
12. Pulse oximetry of > 90% on room air
13. Available multivirus-specific CTLs
14. Negative pregnancy test in female patients if applicable (childbearing potential who have received a reduced intensity conditioning regimen).
15. Written informed consent and/or signed assent line from patient, parent or guardian.

Exclusion Criteria:

1. Patients receiving ATG, or Campath or other immunosuppressive T cell monoclonal antibodies within 28 days of screening for enrollment.
2. Patients with other uncontrolled infections. For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment. For fungal infections patients must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to enrollment.

   Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
3. Patients who have received donor lymphocyte infusion (DLI) within 28 days.
4. Patients with active acute GVHD grades II-IV.
5. Active and uncontrolled relapse of malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-09; Primary Completion 2016-08 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Heslop, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Papadopoulou A, Gerdemann U, Katari UL, Tzannou I, Liu H, Martinez C, Leung K, Carrum G, Gee AP, Vera JF, Krance RA, Brenner MK, Rooney CM, Heslop HE, Leen AM. Activity of broad-spectrum T cells as treatment for AdV, EBV, CMV, BKV, and HHV6 infections after HSCT. Sci Transl Med. 2014 Jun 25;6(242):242ra83. doi: 10.1126/scitranslmed.3008825. PMID 24964991

RESULTS

PARTICIPANT FLOW:
Groups:
- Multivirus-specific T Cells 5*10^6 mCTLs/m2 for Prophylaxis: Cohort 1 prophylaxis: Participants were administrated 5*10^6 mCTLs/m multivirus-specific T cells intravenously for prophylaxis of EBV, CMV, Adenovirus, HHV6 and BK virus infections post allogeneic stem cell transplant.
- Multivirus-specific T Cells 5*10^6 mCTLs/m2 for Treatment: Cohort 1 treatment: Participants were administrated 5*10^6 mCTLs/m multivirus-specific T cells intravenously for treatment of EBV, CMV, Adenovirus, HHV6 and BK virus infections post allogeneic stem cell transplant.
- Multivirus-specific T Cells 1*10^7 mCTLs/m2 for Prophylaxis: Cohort 2 prophylaxis: Participants were administrated 1*10^7 mCTLs/m multivirus-specific T cells intravenously for prophylaxis of EBV, CMV, Adenovirus, HHV6 and BK virus infections post allogeneic stem cell transplant.
- Multivirus-specific T Cells 1*10^7 mCTLs/m2 for Treatment: Cohort 2 treatment: Participants were administrated 1*10^7 mCTLs/m multivirus-specific T cells intravenously for treatment of EBV, CMV, Adenovirus, HHV6 and BK virus infections post allogeneic stem cell transplant.
- Multivirus-specific T Cells 2*10^7 mCTLs/m2 for Prophylaxis: Cohort 3 prophylaxis: Participants were administrated 2*10^7 mCTLs/m multivirus-specific T cells intravenously for prophylaxis of EBV, CMV, Adenovirus, HHV6 and BK virus infections post allogeneic stem cell transplant.
- Multivirus-specific T Cells 2*10^7 mCTLs/m2 for Treatment: Cohort 3 treatment: Participants were administrated 2*10^7 mCTLs/m multivirus-specific T cells intravenously for treatment of EBV, CMV, Adenovirus, HHV6 and BK virus infections post allogeneic stem cell transplant.
Period: Cohort 1: Dose Level 1
Arm/Group | Multivirus-specific T Cells 5*10^6 mCTLs/m2 for Prophylaxis | Multivirus-specific T Cells 5*10^6 mCTLs/m2 for Treatment | Multivirus-specific T Cells 1*10^7 mCTLs/m2 for Prophylaxis | Multivirus-specific T Cells 1*10^7 mCTLs/m2 for Treatment | Multivirus-specific T Cells 2*10^7 mCTLs/m2 for Prophylaxis | Multivirus-specific T Cells 2*10^7 mCTLs/m2 for Treatment
Started | 1 | 3 | 0 | 0 | 0 | 0
Completed | 1 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Received other hematopoietic cells | 0 | 1 | 0 | 0 | 0 | 0
Period: Cohort 2: Dose Level 2
Arm/Group | Multivirus-specific T Cells 5*10^6 mCTLs/m2 for Prophylaxis | Multivirus-specific T Cells 5*10^6 mCTLs/m2 for Treatment | Multivirus-specific T Cells 1*10^7 mCTLs/m2 for Prophylaxis | Multivirus-specific T Cells 1*10^7 mCTLs/m2 for Treatment | Multivirus-specific T Cells 2*10^7 mCTLs/m2 for Prophylaxis | Multivirus-specific T Cells 2*10^7 mCTLs/m2 for Treatment
Started | 0 | 0 | 2 | 2 | 0 | 0
Completed | 0 | 0 | 1 | 1 | 0 | 0
Not Completed | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Received other hematopoietic cells | 0 | 0 | 0 | 1 | 0 | 0
Period: Cohort 3: Dose Level 3
Arm/Group | Multivirus-specific T Cells 5*10^6 mCTLs/m2 for Prophylaxis | Multivirus-specific T Cells 5*10^6 mCTLs/m2 for Treatment | Multivirus-specific T Cells 1*10^7 mCTLs/m2 for Prophylaxis | Multivirus-specific T Cells 1*10^7 mCTLs/m2 for Treatment | Multivirus-specific T Cells 2*10^7 mCTLs/m2 for Prophylaxis | Multivirus-specific T Cells 2*10^7 mCTLs/m2 for Treatment
Started | 0 | 0 | 0 | 0 | 1 | 12
Completed | 0 | 0 | 0 | 0 | 1 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Received other hematopoietic cells | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Eligible patients who received multivirus-specific T cells per protocol.
Groups:
- Multivirus-specific T Cells 5*10^6 mCTLs/m2: Cohort 1 (prophylaxis and treatment): Participants were administrated 5*10^6 mCTLs/m multivirus-specific T cells intravenously for the prophylaxis and treatment of EBV, CMV, Adenovirus, HHV6 and BK virus infections post allogeneic stem cell transplant.
- Multivirus-specific T Cells 1*10^7 mCTLs/m2: Cohort 2 (prophylaxis and treatment): Participants were administrated 1*10^7 mCTLs/m multivirus-specific T cells intravenously for the prophylaxis and treatment of EBV, CMV, Adenovirus, HHV6 and BK virus infections post allogeneic stem cell transplant.
- Multivirus-specific T Cells 2*10^7 mCTLs/m2: Cohort 3 (prophylaxis and treatment): Participants were administrated 2*10^7 mCTLs/m multivirus-specific T cells intravenously for the prophylaxis and treatment of EBV, CMV, Adenovirus, HHV6 and BK virus infections post allogeneic stem cell transplant.
- Total: Total of all reporting groups
Arm/Group | Multivirus-specific T Cells 5*10^6 mCTLs/m2 | Multivirus-specific T Cells 1*10^7 mCTLs/m2 | Multivirus-specific T Cells 2*10^7 mCTLs/m2 | Total
Number analyzed (Participants) | 4 | 4 | 13 | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [9 to 54] | 12 [8 to 17] | 9 [3 to 13] | 9 [6 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5
  Male | 2 | 2 | 12 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 4 | 6 | 12
  African American | 0 | 0 | 2 | 2
  Hispanic or Latino | 2 | 0 | 4 | 6
  Asian | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a DLT
Description: DLT is defined as acute GvHD grades III-IV within 42 days of the last dose of CTLs, # of patients with Grade 3-5 infusion-related adverse events within 30 days of the last dose of CTLs, and # of patients with Grade 4-5 non-hematological adverse events within 30 days of the last dose of CTLs. GVHD grade III-IV scoring is based on the Blood and Marrow Transplant Clinical Trials Network (BMT CTN) GVHD scoring stamp or equivalent. Grade 3-5 infusion-related adverse events and Grade 4-5 non-hematological adverse events are graded by the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 4.X.
Time Frame: 42 days
Population: Data is reported for all participants who received multivirus-specific T cells. A participant is not evaluable for DLT if the participant was removed from the study before 42 days follow up due to a reason other than DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Multivirus-specific T Cells 5*10^6 mCTLs/m2 | Multivirus-specific T Cells 1*10^7 mCTLs/m2 | Multivirus-specific T Cells 2*10^7 mCTLs/m2
Number analyzed (Participants) | 4 | 4 | 13
Participants
  DLT | 0 | 0 | 0
  No DLT | 3 | 4 | 13
  Not evaluable | 1 | 0 | 0

2. Secondary Outcome: Percentage of Patients Who Have a Response in Anti-viral Activity
Description: Percentage of patients who have a response in anti-viral activity that is defined as a viral load reduction to the normal level for at least one of the five virus types
Time Frame: 42 days
Population: Data is reported for all participants who received multivirus-specific CTLs for treatment of EBV, CMV, adenovirus, HHV6 and BK virus.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Multivirus-specific T Cells 5*10^6 mCTLs/m2 for Treatment | Multivirus-specific T Cells 1*10^7 mCTLs/m2 for Treatment | Multivirus-specific T Cells 2*10^7 mCTLs/m2 for Treatment
Number analyzed (Participants) | 3 | 2 | 12
percentage of participants | 66.7 [9.4 to 99.2] | 100 [15.8 to 100] | 83.3 [51.6 to 97.9]

3. Secondary Outcome: Percentage Change of Viral Load From Baseline to Follow-up
Description: Percentage change of viral load by PCR from baseline to follow-up. A positive number indicates a percentage decrease and a negative number indicates a percentage increase.
Time Frame: 3 months
Population: as for outcome 2
Measure: Median (Full Range); unit: percentage change
Groups:
- Multivirus-specific T Cells 1*10^7 mCTLs/m2 for Treatment: Cohort 2 treatment: Participants were administrated 1*10^7 mCTLs/m multivirus-specific T cells intravenously for the prophylaxis and treatment of EBV, CMV, Adenovirus, HHV6 and BK virus infections post allogeneic stem cell transplant.
- Multivirus-specific T Cells 2*10^7 mCTLs/m2 for Treatment: Cohort 3 treatment: Participants were administrated 2*10^7 mCTLs/m multivirus-specific T cells intravenously for the prophylaxis and treatment of EBV, CMV, Adenovirus, HHV6 and BK virus infections post allogeneic stem cell transplant.
Arm/Group | Multivirus-specific T Cells 5*10^6 mCTLs/m2 for Treatment | Multivirus-specific T Cells 1*10^7 mCTLs/m2 for Treatment | Multivirus-specific T Cells 2*10^7 mCTLs/m2 for Treatment
Number analyzed (Participants) | 3 | 2 | 12
percentage change
  Adv: number analyzed (Participants) | 0 | 0 | 3
  Adv |  |  | 100 [100 to 100]
  BKV: number analyzed (Participants) | 2 | 0 | 6
  BKV | 100 [100 to 100] |  | 100 [-27.6 to 100]
  CMV: number analyzed (Participants) | 1 | 1 | 5
  CMV | 99.2 [99.2 to 99.2] | 100 [100 to 100] | 100 [-4.2 to 100]
  EBV: number analyzed (Participants) | 1 | 1 | 1
  EBV | 100 [100 to 100] | 100 [100 to 100] | 100 [100 to 100]
  HHV6: number analyzed (Participants) | 0 | 1 | 2
  HHV6 |  | 100 [100 to 100] | -7.0 [-14.0 to 0]

4. Secondary Outcome: Median Peak Frequency of Specific T Cells Post-infusion
Description: Median peak frequency of specific T cells as measured by Elispot to assess reconstitution of antiviral immunity.
Time Frame: 3 months
Population: as for outcome 2
Measure: Median (Full Range); unit: spot forming cells/5 * 10^5 input cells
Groups:
- Multivirus-specific T Cells 5*10^6 mCTLs/m2 for Treatment: Cohort 1 treatment: Participants were administrated 5*10^6 mCTLs/m multivirus-specific T cells intravenously for the prophylaxis and treatment of EBV, CMV, Adenovirus, HHV6 and BK virus infections post allogeneic stem cell transplant.
Arm/Group | Multivirus-specific T Cells 5*10^6 mCTLs/m2 for Treatment | Multivirus-specific T Cells 1*10^7 mCTLs/m2 for Treatment | Multivirus-specific T Cells 2*10^7 mCTLs/m2 for Treatment
Number analyzed (Participants) | 3 | 2 | 12
spot forming cells/5 * 10^5 input cells
  ADV: number analyzed (Participants) | 0 | 0 | 3
  ADV |  |  | 224.0 [6.0 to 225.0]
  BKV: number analyzed (Participants) | 2 | 0 | 6
  BKV | 42.3 [10.5 to 74.0] |  | 271.3 [5.0 to 932.0]
  CMV: number analyzed (Participants) | 1 | 1 | 5
  CMV | 28.5 [28.5 to 28.5] | 1023.0 [1023.0 to 1023.0] | 884.5 [386.0 to 2656.0]
  EBV: number analyzed (Participants) | 1 | 1 | 1
  EBV | 497.0 [497.0 to 497.0] | 40.0 [40.0 to 40.0] | 224.0 [224.0 to 224.0]
  HHV6: number analyzed (Participants) | 0 | 1 | 2
  HHV6 |  | 175.0 [175.0 to 175.0] | 24.8 [3.0 to 46.5]

ADVERSE EVENTS:
Time Frame: Data on adverse experiences/toxicities regardless of seriousness must be collected for documentation purposes only for 30 days after the last dosing of the study drug/biologic with the exception of acute GVHD which will be followed for 6 weeks.
Arm/Group | Multivirus-specific T Cells 5*10^6 mCTLs/m2 | Multivirus-specific T Cells 1*10^7 mCTLs/m2 | Multivirus-specific T Cells 2*10^7 mCTLs/m2
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/4 | 4/13
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multivirus-specific T Cells 5*10^6 mCTLs/m2 (N=4) | Multivirus-specific T Cells 1*10^7 mCTLs/m2 (N=4) | Multivirus-specific T Cells 2*10^7 mCTLs/m2 (N=13)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (2) | 1 (1)
Infections and infestations - Other, specify: RSV (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify: rhinovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urethral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify: dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify: Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify: lung inflitrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multivirus-specific T Cells 5*10^6 mCTLs/m2 (N=4) | Multivirus-specific T Cells 1*10^7 mCTLs/m2 (N=4) | Multivirus-specific T Cells 2*10^7 mCTLs/m2 (N=13)
Anemia (Blood and lymphatic system disorders) | 4 (25) | 3 (12) | 10 (38)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (4) | 1 (1) | 2 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (10) | 2 (2) | 4 (7)
Gastrointestinal disorders - Other, specify: Intercurrent gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (4) | 1 (1) | 5 (6)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 7 (10)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 7 (8)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 2 (2)
General disorders and administration site conditions - Other, specify: PICC line pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
General disorders and administration site conditions - Other, specify: flank pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify: pain- knees (General disorders) | 0 (0) | 1 (2) | 0 (0)
General disorders and administration site conditions - Other, specify: pain- legs (General disorders) | 0 (0) | 1 (2) | 0 (0)
Irritability (General disorders) | 0 (0) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 2 (3)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify: Rhinovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify: clostridium difficile (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, specify: human herpes virus 7 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, specify: oral thrush (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify: oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Infections and infestations - Other, specify: rhinovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Mucosal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (5)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 2 (2) | 4 (8)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 3 (5)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 3 (7)
Hemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Lymphocyte count decreased (Investigations) | 4 (12) | 1 (1) | 11 (36)
Neutrophil count decreased (Investigations) | 2 (5) | 1 (3) | 9 (45)
Platelet count decreased (Investigations) | 3 (20) | 1 (2) | 8 (56)
White blood cell decreased (Investigations) | 4 (11) | 2 (9) | 10 (39)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (15) | 2 (3) | 8 (27)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (6) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (5)
Hypokalemia (Metabolism and nutrition disorders) | 1 (9) | 1 (1) | 4 (15)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (5) | 0 (0) | 5 (8)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 5 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (7) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify: delayed speech (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify: right hand weakness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (2) | 3 (5)
Proteinuria (Renal and urinary disorders) | 1 (1) | 3 (4) | 3 (6)
Renal and urinary disorders - Other, specify: dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify: rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Purpura (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (5)
Skin and subcutaneous tissue disorders - Other, specify: diaper rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify: lacy rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: umbilical wound (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (4) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No